CLINICAL TRIAL: NCT04155684
Title: Dysbiosis Impact on Lung Disease in HIV
Acronym: DimPL
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alison Morris, Chief, Pulmonary, Allergy, and Critical Care Medicine, University of Pittsburgh
Other Study IDs: STUDY19060360; R01HL138630 (NIH)
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2022-10

CONDITIONS: HIV Infections; COPD; Microbiome
Keywords: microbiome
MeSH Terms: conditions — HIV Infections; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, oral samples, bronchial wash and stool will be stored in Dr. Morris's lab at the University of Pittsburgh indefinitely.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HIV + with COPD: COPD will be defined as Subjects with FEV1/FVC<0.70 or FEV1 and DLco < 80% predicted
- HIV+ normal: Normal PFT's

SUMMARY:
Despite the high burden of respiratory symptoms in the HIV+ population, causes of chronic obstructive pulmonary disease (COPD) in individuals with HIV are poorly understood. Microbial communities present in the lungs or gut could play an important role in COPD via their ability to stimulate inflammation and oxidative stress and by the interactions of microbial and host gene transcription. By exploring the impact of the structure and function of microbial communities on the host in HIV-associated COPD, this project could lead to discovery of novel therapeutics to treat and prevent COPD. Subjects will be 20 HIV+ individuals with COPD (FEV1/FVC <0.70 and FEV1 and DLco<80% predicted) and 20 HIV+ individuals with normal lung function (controls) and 10 HIV negative individuals recruited from our ongoing cohorts. Controls will be matched to the individuals with COPD based on age, gender, pack-years of smoking, ART use, HIV viral suppression, and history of illicit drug use. Bronchoscopy will be performed on all subjects. The investigator will uncover mechanisms that contribute to COPD in HIV+ individuals, which will lead to interventional therapies. For example, the investigators evaluate the impact of bacteria on lung epithelial cell gene expression and inflammation and test ability of anti-inflammatories to alter responses. Identification of other key pathways or microbes could also lead to testing of pro-biotics, post-biotics (bacterial metabolites), or therapy with bacteria genetically modified for desired function or metabolites.

DETAILED DESCRIPTION:
Day one:

Respiratory questionnaires:

The Modified Medical Research Council Dyspnea scale (MMRC) and the St. George's Questionnaire(SGQT) will be administered. These are paper and pencil questionnaires that inquire about respiratory symptoms, quality of life, and other lung related issues. This will take approximately 20 minutes to complete.

Blood Sample collection:

The subject will be asked to provide a blood sample by venipuncture of approximately 110mls (7.4 tablespoon) at this study visit. The purpose of this collection is to have blood processed for serum, plasma, and PBMCS, and a portion stored for RNA to be used for future use. A hemoglobin and carboxyhemoglobin will be done in order to calculate the DLCO only if the participant requires repeat spirometry and DLCO testing. In addition, part of this blood will be used to perform routine clinical blood tests to assure that it is safe to proceed with the bronchoscopy test. (CBC/DIFF/PLT, LYTS, BUN, Creatinine, Glucose, PT/PTT) The de-identified research samples will be processed and stored at -80C. Personal information will not be provided to individual research subjects as Dr. Morris's laboratory is not CLIA certified .

Oral Sample collection:

A one time collection of saliva and tongue scraping will be done at the first visit.

Saliva sample will consist of between 1-5 mL of saliva spit into a sterile collection vessel. Tongue scraping will consist of gentle scraping of the dorsal tongue (not hard enough to cause abrasion) using a blunt, sterile device designed for this purpose that will then be collected in a sterile collection vessel.

Stool collection: The investigator will ask participants to provide a stool sample. They will be instructed on how to collect a stool specimen at home. The investigator will give them instructions and a kit that will provide all the supplies needed to collect the stool and return with it on day 2 of this study.

Lung function testing: (performed if there is not a PFT available from the past 3 months) The routine lung function endpoints of FVC, FEV1, FEV1/FVC, and FEF25-75% will be measured with the flow-volume loop recorder on a NDD Easy One Pro testing system before and after bronchodilator administration. The system is calibrated for body temperature and pressure of saturated gas and volumes, per American Thoracic Society (ATS) standards . DLco will be measured using the automated single-breath procedure of the integrated testing system, which conforms with ATS standards. All testing will be reviewed by (PI). If any concerns or abnormal results are discovered during this testing, a member of the research team will notify the subject or the subject's primary care physician, who will assess the need to provide additional evaluation.

Pregnancy Test: A urine pregnancy test will be performed on all women of child bearing potential. Men and women who are post menopausal for at least 1 year or have been surgically made sterile will not be included.

Day 2: (not necessarily consecutive days but within one week of day 1) Bronchoscopy: Fiber optic bronchoscopy will be performed using the ATS recommendation and institutional protocols for conscious sedation. The testing will be performed by a physician certified in pulmonary medicine and proficient in the procedure and certified by UPMC. Fluoroscopy will not be used. Subjects will be instructed to fast overnight and withhold aspirin and anti-inflammatory analgesics for 48 hours prior to the procedure. Subjects will have undergone a pre- bronchoscopy spirometry within the past 3 months and only clinically stable subjects (FEV1>30% predicted after albuterol) will undergo the procedure. Subjects will also receive Proventil HFA Inhaler 2 puffs, after 5 minutes will receive a second dose of Proventil 2 puffs prior to sending patient to the Bronchoscopy suite. Subjects may receive a drug to dry secretions ( Atropine 0.6mg).

Subjects will receive a local anesthetic to the upper and lower airways and an intravenous sedative and/or analgesic (midazolam; fentanyl). The midazolam dose will not exceed 10mg and/or the fentanyl dose will not exceed 200 micrograms. Lidocaine will not exceed a dose of 9 mg/kg (0.9 cc of 1%/kg) or a maximum dose of 600 mg (60 cc 1%) during the procedure. Subject monitoring will follow the local protocol for conscious/deep sedation. If needed, subjects will receive additional short acting beta agonist. After transoral insertion of the bronchoscope bronchoalveolar lavage will be performed. Blood pressure, heart rate, and oxygen saturation will be monitored throughout the procedure. The physician may stop the procedure at any time for clinical safety.

Bronchoalveolar lavage:

BAL will be performed with room temperature normal saline. After wedging the bronchoscope in a (sub)segmental bronchus, approximately 50cc of saline will be instilled with each washing and withdrawn by syringe aspiration. This will be repeated up to 4 times per segment as needed. Amount of wash and selection of segments will be at the discretion of the physician. Many clinical bronchoscopies are within this range of volume, and research bronchoscopies have been found to be safe with volumes ranging from 100 to 300 cc even in subjects with severe asthma (Wenzel S et al. Bronchoscopic evaluation of severe asthma. American Journal of Respiratory and Critical Care Medicine 1997;156:737-43; Summary and recommendations of a workshop on the investigative use of fiberoptic bronchoscopy and bronchoalveolar lavage in asthmatic patients. Chest 1985;88:136-38). The investigator will stop the lavage at any point where the investigators do not feel that it would be clinically tolerated by the patient.

The volume collected after each withdrawal will be recorded.

Bronchial brushing:

Cytology bronchial brushing involves positioning the bronchoscope at the right middle or lower lobe, passing a cytology brush through the bronchoscope and gently brushing the lining of the airways. This may be repeated at least eight more times per segment to ensure an adequate sample collection. If any sample collected is not acceptable or adequate for analysis, another sample may be collected so long as the physician performing the bronchoscopy procedure decides that no significant risk is present with the additional collection.

1. Participant will be monitored at UPMC Montefiore until the sedation has worn off. After the bronchoscopy is completed, the subject will wait in the bronchoscopy recovery area or the clinical research CTRC to make sure thier breathing has not been affected by the procedure and to be sure that the anesthesia has worn off. Pulse oximetry monitoring will continue throughout recovery period. If the subject is not able to breathe as well as they could before the bronchoscopy, the investigator will give additional albuterol and check the breathing again.Participant will not be allowed to leave the recovery area until their breathing is back to their normal level. If a participants breathing does not return to baseline they will be required to be admitted overnight.
2. Participant will not be allowed to drive themselves home after the bronchoscopy.

Bronchoscopy pre and post sedation care will be conducted in the MUH CTRC. Staff are trained research registered nurses and familiar with post bronchoscopy monitoring. Pulse oximetry will be closely monitored and the subject will not be discharged until anesthesia has worn off and the subject's breathing is back to normal.

The bronchoscopy procedure will take about 45 minutes, the participant will not be discharged until anesthesia has worn off and their breathing is back to normal.

All bronchoscopies will be done in the pulmonary division bronchoscopy suite. Resuscitative equipment and personnel are present in the room to minimize risk.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, documented in medical record at any time prior to study entry.
2. HIV negative who have prior involvement in an HLRC study.
3. Men and women age 18 to 80.
4. Ability and willingness to complete all tests.
5. Participant in HLRC studies,(PRO10060177, PRO09050521, PRO14070355, PRO08030011, PRO00606151, PRO13050229) MACS(Pitt Men's study), Women's Interagency Health Study, PACT or local HIV + clinics.
6. COPD will be defined as Subjects with FEV1/FVC<0.70 or FEV1 and DLco < 80% predicted - this is the same criteria for the other HLRC studies listed in #5.

Exclusion Criteria:

1. Pregnancy or breast-feeding. (urine pregnancy done on all females of child bearing potential-males and females who are at least 1 year post menopausal or surgically sterile will not be tested)
2. Contraindication to pulmonary function testing (i.e. abdominal or cataract surgery within 3 months, recent myocardial infarction, etc.).
3. Increasing respiratory symptoms or febrile (temperature >100.40F [380C]) within 4 weeks of study entry.
4. Acute cardiopulmonary issue in the past 4 months.
5. Uncontrolled hypertension at screening visit (systolic > 180 mm Hg or diastolic > 100 mm Hg) from an average of two or more readings. Subject may return for screening after blood pressure is controlled.
6. Active cancer requiring systemic chemotherapy or radiation.
7. Active infection of lungs, brain, or abdomen.
8. Intravenous drug use or alcohol use that will impair ability to complete study investigations in the opinion of the investigator.
9. subjects with an upper or lower respiratory tract infection
10. Individuals with a Primary diagnosis of vocal cord dysfunction, or those with significant or uncontrolled systemic diseases, for example; uncontrolled diabetes or uncontrolled hypertension.
11. on antibiotics in the past 3 months for an acute infection (prophylaxis OK)
12. FEV1 less than 30% predicted
13. Allergy to any drug needed to perform testing and no alternative available (albuterol, atropine, lidocaine, fentanyl, versed, Demerol)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women HIV positive or HIV negative who have participated in The HIV Lung Research group studies in the past.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Ig-bound and BAL bacteria | 5 years
  Using 16S sequencing, we will compare unsorted bacteria from BAL to IgG- and IgM-bound and Ig-negative bacteria in HIV+ individuals with and without COPD.
AEC supernatant cytokines and cell gene expression | 5 years
  Basolateral supernatant cytokines and MMPs will be measured by ELISA, and AEC cytokine and MMP gene expression by rtPCR. We will determine if IgG- or IgM-bound bacteria from HIV+ individuals with COPD generate a greater inflammatory response in co-culture than bacteria from HIV+ individuals without COPD and if this response can be decreased by anti-inflammatories.
AEC function | 5 years
  Trans-epithelial electrical resistance (TEER) will be measured hourly during bacterial co-culture with ALI AECs in the various experimental conditions using an Ag/AgCl electrode106

CONTACTS AND LOCATIONS:
Overall Officials: Alison J Morris, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburagh, Pittsburgh, Pennsylvania, United States